CLINICAL TRIAL: NCT06064461
Title: Vitaccess Real MG Registry: A Prospective International Observational Patient Registry in Myasthenia Gravis Linking Clinical and Patient-reported Data.
Brief Title: Vitaccess Real MG Registry
Acronym: VRMG
Status: Recruiting | Type: Observational
Sponsor: Vitaccess Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 5137-Vitaccess-MG-01
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; patient registry; longitudinal; observational data
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Vitaccess Real MG (VRMG) is a patient registry designed to capture longitudinal observational data on myasthenia gravis (MG), its treatment, and impact on symptoms, daily activities, and quality of life (QoL). The duration of the registry is 10 years from launch, and approximately 600 patients will be recruited in the US and Europe with no defined upper limit. The registry will link relevant patient- and healthcare professional (HCP)-reported data with clinical data from medical records.

Patients will be recruited at clinical sites in all participating countries. In the US only, patients can additionally be recruited via community neurologists or direct-to-patient recruitment.

DETAILED DESCRIPTION:
Traditional site recruitment (all countries):

Adult patients who are being treated for MG at one of the participating clinics or centers in one of the participating countries (currently the US and UK) at the time of enrolment and who meet the inclusion and exclusion criteria will be identified and approached by their clinical team and invited to participate in the registry.

Patient-reported data will be collected via the VRMG Registry platform, a digital data capture platform accessible via any web-enabled platform (e.g., phone, tablet, laptop, computer). Custom survey and patient-reported outcomes data will be collected at baseline and at regular intervals thereafter for a follow-up period of up to 10 years. The data collected will capture the impact of MG on daily living, fatigue, and health-related quality of life.

Site research teams will complete and update an eCRF (every six months ± one months) for each patient, including data from the patient's EMR. eCRFs that are completed within one months prior to or following each six-month mark will be considered within the same assessment window for analytics purposes so that patients will not be required to visit the clinical site for the purposes of the registry outside of their regular clinical visits.

Community neurologist recruitment (US only):

Community neurologists who are treating MG patients who would be eligible for participation in the registry will be able to register their interest for involvement and provide details of their credentials via an informational website. Approved community neurologists will identify and approach potential participants, who will participate in the registry as normal. Clinical data will be captured from participants' electronic medical records via an EMR aggregator.

Direct-to-patient recruitment (US only):

A cohort of US-based participants in the MyRealWorld MG study - a longitudinal observational study in MG that Vitaccess has run since 2019 - have provided consent to be contacted by Vitaccess about future research. Vitaccess will contact this patient cohort directly via email to introduce them to the registry; patients can access the registry's informational website to get further information. Clinical data will be captured from participants' electronic medical records via an EMR aggregator.

Patient-reported and eCRF data will be linked via a unique ID and PIN assigned to each participant at enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years) with a clinically-confirmed diagnosis of myasthenia gravis (MG).
* Resident in one of the scope countries.
* Access to a smartphone/tablet/computer/laptop
* Willing and able to provide informed consent in their local language to take part in the study.

Exclusion Criteria:

* Participation in a clinical trial at the time of study enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are being treated for MG at one of the participating clinics or centers in one of the study countries at the time of enrolment and who meet the inclusion and exclusion criteria will be identified and approached by their clinical team and invited to participate in the registry.
  Adult patients in the US who are not being treated at a participating clinic will be able to enrol via their community neurologist or direct-to-patient recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2034-07 (Estimated); Study Completion 2034-07 (Estimated)

PRIMARY OUTCOMES:
The Vitaccess Real MG Registry | 10 years
  A patient registry designed to capture longitudinal observational data on myasthenia gravis (MG), its treatment, and impact on symptoms, daily activities, and quality of life.

SECONDARY OUTCOMES:
Describe the demographic characteristics of patients | At baseline
  EMR data reported by HCPs or captured via EMR aggregator ("Registration Form")
Describe change in clinical trial participation of patients | At follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregator ("Clinical Trial Participation Form")
Describe the diagnosis (date, tests, and symptoms) of patients | At baseline
  EMR data reported by HCPs or captured via EMR aggregator ("Diagnosis Information Form")
Describe change in clinical characteristics of patients. | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregator ("Clinical Characteristics Form")
Describe change in medical history of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregator ("Medical History Form")
Describe change in concomitant treatments received by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregator ("Concomitant Medication Log")
Describe change in routine MG treatments received by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregator ("Routine MG Treatments Log")
Describe change in rescue MG treatments received by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregator ("Rescue MG Treatments Log")
Describe change in severity of MG symptoms experienced by patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  Myasthenia Gravis Activities of Daily Living (MG-ADL) data reported by HCPs or captured via EMR aggregator ("MG-ADL")
Describe change in healthcare resource use of patients | At baseline visit and at follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregator ("Healthcare Resource Use")
Describe change in type and severity of adverse events experienced by patients | At follow-up visits (every 6±1 months) for up to 10 years
  EMR data reported by HCPs or captured via EMR aggregator ("Adverse Events")
Describe change in severity of MG symptoms experienced by patients | At baseline and every 1 month thereafter for up to 10 years.
  Myasthenia Gravis Activities of Daily Living (MG-ADL) data reported by patients via the Vitaccess Real MG Registry platform ("MG-ADL")
Describe change in type and severity of fatigue experienced by patients | At baseline and every 2 months thereafter for up to 10 years.
  MG Symptoms PRO Fatigue Component data reported by patients via the Vitaccess Real MG Registry platform ("MG Symptoms PRO Fatigue Component")
Describe change in type and severity of fatigue experienced by patients | At baseline and every 2 months thereafter for up to 10 years.
  NeuroQoL Fatigue Short Form data reported by patients via the Vitaccess Real MG Registry platform ("NeuroQoL Fatigue Short Form")
Describe change in impact of MG on health-related quality of life of patients | At baseline and every 2 months thereafter for up to 10 years.
  Myasthenia Gravis Quality of Life 15-item revised scale (MG-QoL-15r) data reported by patients via the Vitaccess Real MG Registry platform ("MG-QoL-15r")

CONTACTS AND LOCATIONS:
Overall Officials: Mark JW Larkin, PhD, Principal Investigator — Vitaccess Ltd
Locations (8):
- United States (6):
  - UCI Health, Orange, California
  - HSHS St. Elizabeth's Hospital, O'Fallon, Illinois
  - UK HealthCare - University of Kentucky, Lexington, Kentucky
  - Neurology Associates of South Jersey, Lumberton, New Jersey
  - Medical University South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center at Houston, Houston, Texas
- United Kingdom (2):
  - Vitaccess Ltd, London, London
  - University Hospitals Birmingham, Birmingham

IPD SHARING:
Plan to Share IPD: No